CLINICAL TRIAL: NCT04465864
Title: Randomized, Controlled Treatment With an Intracanalicular Dexamethasone (0.4mg) Insert Following Cataract Surgery With IOL Combined With MIGS, Specifically iStent, iStent Inject or KDB in Patients With POAG or Ocular Hypertension (OHTN)
Brief Title: Investigate, Following Cataract Surgery With IOL in Conjunction With Intracanalicular Dexamethasone Insert
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wolstan and Goldberg Eye Associates (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEXTENZA
Record Dates: First submitted 2020-02-12; First posted 2020-07-10 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Glaucoma, Primary Open Angle; Cataract
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract | interventions — Mutagenesis, Insertional; Drug Implants

STUDY DESIGN:
Intervention Model Description: Group 1: intracanalicular dexamethasone (0.4 mg) insertion four days (+/- 1 day) prior to cataract surgery with intraocular lens (IOL) implant and MIGS (iStent, iStent inject or KDB) insertion. (Patient to use antibiotic three days prior to surgery)
  Group 2: intracanalicular dexamethasone (0.4 mg) insertion on the day of cataract surgery with intraocular lens (IOL) implant and MIGS (iStent, iStent inject or KDB) insertion. (Patient to use antibiotic three days prior to surgery)
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insertion visit 4 days prior (Other): Intracanalicular dexamethasone (0.4 mg) insertion four days (+/- 1 day) prior to cataract surgery with intraocular lens (IOL) implant and MIGS (iStent, iStent inject or KDB) insertion. (Patient to use antibiotic three days prior to surgery)
  Interventions: Drug: Intracanalicular Dexamethasone, 0.4 mg insert
- Surgical 1 visit day 0 (Other): Intracanalicular dexamethasone (0.4 mg) insertion on the day of cataract surgery with intraocular lens (IOL) implant and MIGS (iStent, iStent inject or KDB) insertion. (Patient to use antibiotic three days prior to surgery)
  Interventions: Drug: Intracanalicular Dexamethasone, 0.4 mg insert

INTERVENTIONS:
Drug: Intracanalicular Dexamethasone, 0.4 mg insert — Intracanalicular Dexamethasone, 0.4 mg insert four days (+/- 1 day) prior to surgery or inserted the day of surgery.
  Other Names: MIGS (iStent, iStent inject or KDB) insertion.

SUMMARY:
Randomized, controlled treatment with an intracanalicular dexamethasone (0.4mg) insert following cataract surgery with intraocular lens implant (IOL) combined with minimally invasive glaucoma surgery (MIGS), specifically iStent, iStent inject or KDB in patients with primary open angle glaucoma (POAG) or ocular hypertension (OHTN)

DETAILED DESCRIPTION:
To determine treatment and patient reported outcomes, following cataract surgery with intraocular lens implant in conjunction with minimally invasive glaucoma surgery (MIGS) more specifically iStent, iStent inject or KDB with an intracanalicular dexamethasone (0.4 mg) insert, inserted four days (+/- 1 day) prior to surgery as compared to insertion on day of surgery. Patients with either primary open angle glaucoma (POAG) or ocular hypertension (OHTN) requiring cataract surgery with IOL implant, will be separated into two groups.

Group 1: intracanalicular dexamethasone (0.4 mg) insertion four days (+/- 1 day) prior to cataract surgery with intraocular lens (IOL) implant and MIGS (iStent, iStent inject or KDB) insertion. (Patient to use antibiotic three days prior to surgery) Group 2: intracanalicular dexamethasone (0.4 mg) insertion on the day of cataract surgery with intraocular lens (IOL) implant and MIGS (iStent, iStent inject or KDB) insertion. (Patient to use antibiotic three days prior to surgery)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Been diagnosed with POAG or OHTN and MIGS (iStent, iStent inject or KDB) has been planned
* Unilateral or bilateral cataract surgery with IOL has been planned
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria:

* Patients under the age of 18.
* Pregnancy (must be ruled out in women of child-bearing age with pregnancy test)
* Active infectious systemic disease
* Active infectious ocular or extraocular disease
* Unobstructed nasolacrimal duct in the study eye(s)
* Hypersensitivity to dexamethasone
* Patients being treated with immunomodulating agents in the study eye(s)
* History of prior ocular surgery, including Lasik or PRK
* History of ocular inflammation or macular edema
* Patients being treated with >375mg daily of NSAIDs

  o Patients on doses higher than 375mg of oral NSAIDs will be considered if they discontinue the medication 2 weeks prior to the study start date.
* Patients taking inconsistent varying doses of an NSAID on a daily basis.
* Patients being treated with immunosuppressants and/or oral steroids
* Patients with a corticosteroid implant (i.e. Ozurdex)
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Intracanalicular Dexamethasone, 0.4 mg insert four days (+/- 1 day) prior to surgery | four days (+/- 1 day) prior to surgery with visits scheduled at day 1, day 7, day 14, day 30, and day 45.
  Primary: Will receive the insert four days (+/- 1 day) prior to surgery. Each enrolled subject will be required to complete seven scheduled visits over the course of the study period: Baseline, insertion visit, operative visit, Day 1, 7, 30, and a 14 & 45-day phone call.
  Absence of cells in anterior chamber at day 7 as measured by: Summed Ocular Inflammation Score (0-4) Absence of cell to be defined as a grade of (0-0.5) Absence of pain at Day 7 (score of 0) as measured by ocular pain assessment numerical grading scale 0-10 Mean change in BCVA from baseline (Day 7,30) Mean change in OCT from baseline (Day 30) Physician ease of intracanalicular insertion evaluation as measured by physician questionnaire Incidence and severity of ocular and systemic AE's (Day 1,7,14,30,45)

SECONDARY OUTCOMES:
Intracanalicular Dexamethasone, 0.4 mg insertion on day of surgery. | insertion on day of surgery with scheduled visits on day 1, day 7, day 14, day 30, and day 45.
  Secondary: Will receive the insert on the day of surgery. Each enrolled study subject will be required to complete six scheduled visits over the course of the study period: Screening visit, operative/insertion visit, Day 1, 7, 30, and a 14 & 45 day phone call.
  Measuring cell, pain and flare at (Day 1,30) Absence of cell to be defined as a grade of (0-0.5) Absence of flare to be defined as a grade of (0-1) Determining if call backs have decreased at the clinic with study patients

CONTACTS AND LOCATIONS:
Overall Officials: Damien Goldberg, MD, Principal Investigator — Wolstan & Goldberg Eye Associates
Locations (1):
- Wolstan and Goldberg Eye Associates, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No